CLINICAL TRIAL: NCT02627963
Title: A Phase 3, Randomized, Controlled, Multi-Center, Open-Label Study to Compare Tivozanib Hydrochloride to Sorafenib in Subjects With Refractory Advanced Renal Cell Carcinoma
Brief Title: A Study to Compare Tivozanib Hydrochloride to Sorafenib in Participants With Refractory Advanced Renal Cell Carcinoma (RCC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AV-951-15-303
Record Dates: First submitted 2015-12-09; First posted 2015-12-11 (Estimated); Results first posted 2020-02-20 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-06

CONDITIONS: Carcinoma, Renal Cell
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tivozanib hydrochloride (Experimental): Participants randomized to this arm will receive the study drug, tivozanib hydrochloride.
  Interventions: Drug: Tivozanib hydrochloride
- Sorafenib (Active Comparator): Participants randomized to this arm will receive the comparator drug, sorafenib.
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Tivozanib hydrochloride — Tivozanib hydrochloride
  Arms: Tivozanib hydrochloride
Drug: Sorafenib — Sorafenib
  Arms: Sorafenib

SUMMARY:
This is a Phase 3, open-label, randomized, controlled, multi-national, multi-center, parallel-arm study comparing tivozanib to sorafenib in participants with refractory advanced renal cell carcinoma (RCC).

Participants will be randomized (1:1) to treatment with tivozanib or sorafenib.

Participants will be stratified by International Metastatic Renal Cell Carcinoma Database Consortium (IMDC) risk category (favorable; intermediate; poor) and prior therapy (two prior vascular endothelial growth factor receptor tyrosine kinase inhibitors (VEGFR TKI); a prior checkpoint inhibitor [programmed cell death -1 protein (PD-1) or PD-1 ligand (PD1-L) inhibitor] plus a prior VEGFR TKI; a prior VEGFR TKI plus any other systemic agent).

All participants will be evaluated for progression free survival, overall survival, objective response rate, and the duration of response as well as safety and tolerability.

Pharmacokinetic (PK) analyses are also included in study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Participants with metastatic RCC who have failed 2 or 3 prior systemic regimens, one of which includes a VEGFR TKI other than sorafenib or tivozanib.
* Histologically or cytologically confirmed RCC with a clear cell component (participants with pure papillary cell tumor or other non-clear cell histologies, including collecting duct, medullary, chromophobe, and unclassified RCC are excluded).
* Measurable disease per the Response Evaluation Criteria in Solid Tumors (RECIST) criteria Version 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy ≥ 3 months.

Exclusion Criteria:

* Prior treatment with sorafenib or tivozanib.
* More than 3 prior regimens for metastatic RCC.
* Known central nervous system (CNS) metastases other than stable, treated brain metastases. Participants with previously treated brain metastasis will be allowed if the brain metastasis has been stable by neuroimaging without steroid treatment for at least 3 months following prior treatment (radiotherapy or surgery).
* Significant hematologic, gastrointestinal, thromboembolic, vascular, bleeding, or coagulation disorders.
* Significant serum chemistry abnormalities
* Significant cardiovascular disease, including: Active clinically symptomatic left ventricular failure, uncontrolled hypertension, myocardial infarction, severe angina, or unstable angina within 6 months prior to administration of first dose of study drug, history of serious ventricular arrhythmia, cardiac arrhythmias requiring anti-arrhythmic medications.
* Inadequate recovery from any prior surgical procedure or major surgical procedure within 4 weeks prior to administration of first dose of study drug.
* Currently active second primary malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2016-05-24 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2021-06-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (190):
- United States (56):
  - University Of UA Cancer Center(UACC)/DH-SJHMC, Phoenix, Arizona
  - Arizona Oncology Associates, PC - HAL, Phoenix, Arizona
  - Arizona Oncology - Phoenix - Deer Valley Women's Center Loca, Phoenix, Arizona
  - Arizona Oncology - Scottsdale, Scottsdale, Arizona
  - City of Hope Comprehensive Breast Cancer Center, Duarte, California
  - Long Beach Memorial Medical Center, Fountain Valley, California
  - Marin Cancer Care, Greenbrae, California
  - UCLA, Los Angeles, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Loyola University Medical Center, Maywood, Illinois
  - Investigative Clinical Research of Indiana, Indianapolis, Indiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Midwest Cancer Center, Omaha, Nebraska
  - Urology Cancer Center, PC, Omaha, Nebraska
  - Comprehensive Cancer Center Of Nevada, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Comprehensive Cancer Center Of Nevada, Las Vegas, Nevada
  - Comprehensive Cancer Center of Nevada, Las Vegas, Nevada
  - Hackensack University Medical Center - John Theurer Cancer, Hackensack, New Jersey
  - New York Oncology Hematology, P.C., Albany, New York
  - New York Oncology Hematology, PC, Albany, New York
  - New York Oncology Hematology, P.C., Clifton Park, New York
  - New York Presbyterian Hospital, New York, New York
  - Columbia University Medical Center - Herbert Irving Pavilion, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Wake Forest University Baptist Medical Center (WFUBMC), Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio Cancer Specialists, Mansfield, Ohio
  - North Coast Cancer Care, Inc, Sandusky, Ohio
  - Wooster Specialty and Surgery Center, Wooster, Ohio
  - St. Luke University Health Network, Easton, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - Texas Oncology - Austin Midtown, Austin, Texas
  - Texas Oncology-Central Austin Cancer Center, Austin, Texas
  - Texas Oncology - South Austin Cancer Center, Austin, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - Fort Worth 12th Ave, Fort Worth, Texas
  - Texas Oncology SW Fort Worth Cancer Center, Fort Worth, Texas
  - Arizona Oncology Associates, PC - HAL, Fort Worth, Texas
  - Comprehensive Cancer Centers of Nevada (CCCN), Fort Worth, Texas
  - Comprehensive Cancer Centers of Nevada, Fort Worth, Texas
  - Nebraska Cancer Specialists (NCS) - Midwest Cancer Center, Fort Worth, Texas
  - Texas Oncology - El Paso Cancer Treatment Center, Fort Worth, Texas
  - Texas Oncology-El Paso Cancer Treatment Center, Fort Worth, Texas
  - Texas Oncology-Garland, Garland, Texas
  - Baylor College of Medicine - Baylor Clinic, Houston, Texas
  - Texas Oncology - Longview Cancer Center, Longview, Texas
  - Texas Oncology, P.A., Plano, Texas
  - Texas Oncology - Tyler, Tyler, Texas
- Belgium (8):
  - UZ Antwerpen, Edegem, Antwerpen
  - Institut Jules Bordet, Brussels, Brussels Capital
  - Grand Hôpital de Charleroi - Site Notre-Dame, Charleroi, Hainaut
  - CHU Ambroise Paré, Mons, Hainaut
  - Jessa Ziekenhuis - Campus Virga Jesse, Hasselt, Limburg
  - CHU Dinant Godinne UCL Namur, Yvoir, Namur
  - UZ Gent, Ghent, Oost-Vlaanderen
  - AZ Sint-Jan Brugge - Oostende - Campus Sint-Jan, Bruges, West-Vlaanderen
- Canada (4):
  - British Columbia Cancer Agency (BCCA), Vancouver, British Columbia
  - Dr. Leon Richard Oncology Centre, Moncton, New Brunswick
  - London Health Sciences Center, London, Ontario
  - Sunnybrook, Toronto, Ontario
- Czechia (5):
  - Masarykuv onkologicky ustav, Brno, Brno-město
  - FN Hradec Kralove, Hradec Králové, Královéhradecký kraj
  - Fakultni nemocnice Olomouc, Olomouc, Olomoucký kraj
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Fakultni nemocnice v Motole, Prague
- Denmark (3):
  - Herlev Hospital, Herlev, Capital
  - Aarhus Universitetshospital, Aarhus C, Central Jutland
  - Odense Universitetshospital, Odense, Region Syddanmark
- France (11):
  - Hopital Saint-André, Bordeaux, Gironde
  - centre Oscar Lambret, Lille, Hauts-de-France
  - CHRU de Tours - Hopital Bretonneau TOURS, Tours, Indre-et-Loire
  - Institut de Cancérologie de l'Ouest Site Paul Papin, Angers, Maine-et-Loire
  - Institut de cancérologie de Lorraine, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Clinique Victor Hugo, Le Mans, Pays de la Loire Region
  - Institut de Cancerologie de la Loire, Saint-Priest-en-Jarez, Pays de la Loire Region
  - Institut Paoli-Calmettes, Marseille
  - Chu De Poitiers, Poitiers
  - ICO, Saint-Herblain
  - Institut Gustave Roussy, Villejuif
- Germany (15):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Univesitaetsklinik Heidelberg, Heidelberg, Baden-Wurttemberg
  - Kliniken Nordoberpfalz AG, Klinikum Weiden, Weiden, Bavaria
  - Johann Wolfgang Goethe Universität, Frankfurt am Main, Hesse
  - Evangelisches Krankenhaus Bielefeld, Bielefeld, North Rhine-Westphalia
  - SZB Study Center University Hospital Bonn, Bonn, North Rhine-Westphalia
  - Uniklinik Köln Klinik und Poliklinik für Urologie, Cologne, North Rhine-Westphalia
  - Universitätsklinikum des Saarlandes, Homburg, Saarland
  - Universitätsklinikum Carl Gustav Carus, Dresden, Saxony
  - Jena University Hospital, Jena, Thuringia
  - Universitätsklinikum Aachen, Aachen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinikum Muenster, Münster
  - Universität Tübingen, Tübingen
- Hungary (13):
  - Pécsi Tudományegyetem Klinikai Központ, Pécs, Baranya
  - Békés Megyei Pándy Kálmán Kórház, Gyula, Bekes County
  - Borsod-Abaúj-Zemplén Megyei Kórház és Egyetemi Oktató Kórház, Miskolc, Borsod-Abauj Zemplen county
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpo, Szeged, Csongrád megye
  - Debreceni Egyetem Klinikai Központ, Debrecen, Hajdú-Bihar
  - Szent Margit Kórház, Budapest
  - Magyar Honvédség Egészségügyi Központ, Budapest
  - Semmelweis Egyetem, Budapest
  - Országos Onkológiai Intézet, Budapest
  - Egyesített Szent István és Szent László Kórház-Rendelőintéze, Budapest
  - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár
  - Markusovszky Egyetemi Oktatókórház, Szombathely
  - Zala Megyei Korhaz, Zalaegerszeg
- Italy (23):
  - Casa Sollievo della Sofferenza, IRCCS, San Giovanni Rotondo, Foggia
  - Irccs Irst, Meldola, Forli
  - Istituto Clinico Humanitas Rozzano, IRCCS, Rozzano, Milano
  - Usl 7 Siena - Ospedale Alta Valdelsa ASL TOSCANA SUD-EST, Poggibonsi, Siena
  - Istituto di Candiolo, IRCCS, Candiolo, Torino
  - Ospedale S.Donato, AUSL 8 di Arezzo, Arezzo
  - Centro di Riferimento Oncologico IRCCS, Aviano
  - AO Spedali Civili di Brescia, PO Spedali Civili, Brescia
  - P.O. Ss. Annunziata, Chieti
  - ASST-Istituti Ospitalieri di Cremona, AO di Cremona, Cremona
  - AOU Careggi, Florence
  - IRCCS AOU San Martino-IST Istituto Nazionale per la Ricerca, Genova
  - Ospedale Vito Fazzi, ASL Lecce, Lecce
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Ieo, Irccs, Milan
  - AOU Policlinico di Modena, Modena
  - IRCCS Fondazione "Giovanni Pascale", Napoli
  - Istituto Oncologico Veneto IOV-IRCCS, Padua
  - IRCCS Policlinico San Matteo, Pavia
  - PU Campus Bio-medico di Roma, Roma
  - Regina Elena, Istituto Nazionale dei Tumori, IFO, IRCCS, Roma
  - Azienda Ospedaliera San Camillo Forlanini, Roma
  - Azienda Ospedaliera S. Maria di Terni, Terni
- Poland (7):
  - Europejskie Centrum Zdrowia Otwock, Szpital im. F. Chopina, Otwock, Masovian Voivodeship
  - Centrum Onkologii - Instytut im. Marii Sklodowskiej - Curie, Warsaw, Masovian Voivodeship
  - MAGODENT Sp. z o.o. Szpital Onkologiczno-Kardiologiczny, Warsaw, Masovian Voivodeship
  - Szpital Specjalist w Brzozowie Podkarpacki Ośrodek Onkologiczny, Brzozów
  - COPERNICUS Podmiot Leczn. Sp z o.o.,Wojew. Centrum Onkologii, Gdansk
  - NZOZ Vesalius Sp. z o.o., Krakow
  - Uniwersytecki Szpital Kliniczny im. J. Mikulicza-Radeckiego, Wroclaw
- Spain (28):
  - H.G.U. de Elche, Elche, Alicante
  - H.U.Son Espases, Palma, Balearic Islands
  - Institut Català d'Oncologia-Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Institut Catalá d´Oncología (I.C.O.), L'Hospitalet de Llobregat, Barcelona
  - C.S. Parc Taulí, Sabadell, Barcelona
  - H.U.F. Alcorcón, Alcorcón, Madrid
  - H.U.P Hierro-Majadahonda, Majadahonda, Madrid
  - C.H. de Navarra, Pamplona, Navarre
  - H.del Mar, Barcelona
  - H.Sta.Creu i St.Pau, Barcelona
  - H.U.Vall d'Hebrón, Barcelona
  - H. Clinic de Barcelona, Barcelona
  - H.U. Reina Sofía, Córdoba
  - ICO-H.U.Dr.J.Trueta, Girona
  - C.H. de Jaén, Jaén
  - H.G.U. G. Marañón, Madrid
  - H.U. Infanta Leonor, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - H.C. S.Carlos, Madrid
  - H.U. F. Jiménez Díaz, Madrid
  - H.U. 12 de Octubre, Madrid
  - H.U. La Paz, Madrid
  - H. Madrid Norte Sanchinarro, Madrid
  - H.U. Virgen de la Victoria, Málaga
  - H.U.V. Macarena, Seville
  - F.I. Valenciano de Oncología, Valencia
  - H.U.P.La Fe, Valencia
  - H.U. Miguel Servet, Zaragoza
- United Kingdom (17):
  - Addenbrooke's Hospital, Cambridge, Cambridgeshire
  - Beatson West Of Scotland Cancer Centre, Glasgow, Glasgow City
  - Cheltenham General Hospital, Cheltenham, Gloucestershire
  - Southampton University Hospitals Nhs Trust, Southampton, Hampshire
  - East Lancashire Hospitals NHS Trust, Blackburn, Lancashire
  - Lancashire Teaching Hospitals NHS Foundation Trust, Preston, Lancashire
  - Royal Stroke Center, Stoke-on-Trent, Staffordshire
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - St James's University Hospital / Leeds Teaching Hospitals, Leeds
  - The Royal Marsden NHS Foundation Trust, London
  - Charing Cross Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Mount Vernon Cancer Care, Middlesex
  - Nottingham University Hospitals NHS Trust - City Hospital, Nottingham
  - Churchill Hospital [Oncology], Oxford
  - Singleton Hospital, Swansea
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Meza L, McDermott DF, Escudier B, Hutson TE, Porta C, Verzoni E, Atkins MB, Kasturi V, Pal SK, Rini B. Tivozanib in Patients with Advanced Renal Cell Carcinoma Previously Treated With Axitinib: Subgroup Analysis from TIVO-3. Oncologist. 2023 Mar 17;28(3):e167-e170. doi: 10.1093/oncolo/oyac255. PMID 36576430
- [Derived] Szarek M, Needle MN, Rini BI, Pal SK, McDermott DF, Atkins MB, Hutson TE, Escudier BJ. Q-TWiST Analysis of Tivozanib Versus Sorafenib in Patients With Advanced Renal Cell Carcinoma in the TIVO-3 Study. Clin Genitourin Cancer. 2021 Oct;19(5):468.e1-468.e5. doi: 10.1016/j.clgc.2021.03.018. Epub 2021 Apr 3. PMID 33980467
- [Derived] Rini BI, Pal SK, Escudier BJ, Atkins MB, Hutson TE, Porta C, Verzoni E, Needle MN, McDermott DF. Tivozanib versus sorafenib in patients with advanced renal cell carcinoma (TIVO-3): a phase 3, multicentre, randomised, controlled, open-label study. Lancet Oncol. 2020 Jan;21(1):95-104. doi: 10.1016/S1470-2045(19)30735-1. Epub 2019 Dec 3. PMID 31810797

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 350 participants were randomised and 343 were treated.
Groups:
- Tivozanib Hydrochloride: Participants randomized to this arm received the study drug, tivozanib hydrochloride.
- Sorafenib: Participants randomized to this arm received the comparator drug, sorafenib.
Period: Overall Study
Arm/Group | Tivozanib Hydrochloride | Sorafenib
Started | 175 | 175
Completed | 173 | 169
Not Completed | 2 | 6
Not completed — Randomized but not treated | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tivozanib Hydrochloride | Sorafenib | Total
Number analyzed (Participants) | 175 | 175 | 350
Age, Continuous [Median (Full Range); unit: Years] | 62 [34 to 88] | 63 [30 to 90] | 63 [30 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 47 | 96
  Male | 126 | 128 | 254
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 165 | 167 | 332
  Race: Non-white | 10 | 8 | 18
Previous therapies [Count of Participants; unit: Participants]
  Two VEGFR TKIs | 79 | 80 | 159
  Checkpoint inhibitor plus VEGFR TKI | 47 | 44 | 91
  VEGFR TKI plus other systemic agent | 49 | 51 | 100
IMDC risk category [Count of Participants; unit: Participants]
  Favourable | 34 | 36 | 70
  Intermediate | 109 | 105 | 214
  Poor | 32 | 34 | 66

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: The PFS, as assessed by a blinded independent radiological review (IRR), is defined as the time from randomization to first documentation of objective tumor progression (progressive disease) or death due to any reasons whichever comes first. Disease progression per RECIST 1.1 criteria is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first. Disease progression was assessed every 8 weeks (up to approximately 5 years)
Population: Intent-to-treat (ITT) Population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tivozanib Hydrochloride | Sorafenib
Number analyzed (Participants) | 175 | 175
Months | 5.59 [5.29 to 7.33] | 3.88 [3.71 to 5.55]
Statistical Analysis 1: Comparison: Tivozanib Hydrochloride vs Sorafenib; Test type: Superiority; p = 0.0165, Log Rank — A one-sided, log-rank test stratified for IMDC risk category and prior therapy (two VEGFR TKIs vs. a checkpoint inhibitor plus a VEGFR TKI vs. a VEGFR TKI plus any other systemic agent) at a significance level of α = 0.025 was used; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.56 to 0.94]

2. Secondary Outcome: Overall Survival (OS)
Description: The OS is defined as the time from the date of randomization to date of death due to any cause.
Time Frame: Date of randomization to date of death (up to approximately 5 years)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tivozanib Hydrochloride | Sorafenib
Number analyzed (Participants) | 175 | 175
Months | 16.39 [13.44 to 22.21] | 19.15 [14.95 to 24.21]
Statistical Analysis 1: Comparison: Tivozanib Hydrochloride vs Sorafenib; Test type: Superiority; p = 0.8174, Log Rank; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.75 to 1.25]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: The ORR is defined as the percentage of participants who have at least a 30% reduction in the sum of diameters per RECIST (Version 1.1).
Time Frame: Every 8 weeks from date of randomization until disease progression (up to approximately 5 years)
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Tivozanib Hydrochloride | Sorafenib
Number analyzed (Participants) | 175 | 175
Participants | 31 | 14

4. Secondary Outcome: Duration of Response (DOR)
Description: The DOR is defined as the time from the first documentation of objective tumor response to the first documentation of tumor progression per RECIST 1.1 or to death due to any cause.
Time Frame: Assessed every 8 weeks from date of randomization until date of progression (up to approximately 5 years)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tivozanib Hydrochloride | Sorafenib
Number analyzed (Participants) | 175 | 175
Months | NA [12.91 to NA] — The median and upper limit of the 95% confidence interval were not calculable because an insufficient number of participants reached the event. | 5.65 [5.55 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event.

ADVERSE EVENTS:
Time Frame: From first dose to last dose plus 30 days (up to approximately 5 years)
Description: Serious treatment-emergent adverse events and other (non-serious) treatment-emergent adverse events in Safety Population (all participants who received at least 1 dose of study drug) are reported.
Arm/Group | Tivozanib Hydrochloride | Sorafenib
All-Cause Mortality (participants affected / at risk) | 114/175 | 113/175
Serious Adverse Events (participants affected / at risk) | 81/173 | 67/170
Other Adverse Events (participants affected / at risk) | 171/173 | 170/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tivozanib Hydrochloride (N=173) | Sorafenib (N=170)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchial ulceration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 6 | 6
Urinary tract infection (Infections and infestations) | 3 | 1
Influenza (Infections and infestations) | 2 | 0
Appendicitis (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Meningitis aseptic (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Lung abscess (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 4 | 1
Ischaemic stroke (Nervous system disorders) | 2 | 0
Peripheral motor neuropathy (Nervous system disorders) | 2 | 0
Spinal cord compression (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Altered state of consciousness (Nervous system disorders) | 1 | 0
Brain compression (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Paralysis (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Coma (Nervous system disorders) | 0 | 1
Frontal lobe epilepsy (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Optic neuritis (Nervous system disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Anal ulcer (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 3 | 2
Pyrexia (General disorders) | 2 | 1
Death (General disorders) | 1 | 3
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 1
Performance status decreased (General disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatobiliary disease (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Confusional state (Psychiatric disorders) | 3 | 0
Depression (Psychiatric disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 0
Renal failure (Renal and urinary disorders) | 1 | 2
Haematuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 5
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Coronary artery disease (Cardiac disorders) | 0 | 2
Atrial flutter (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Hypertension (Vascular disorders) | 2 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Hypercalcaemia of malignancy (Endocrine disorders) | 2 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Rash morbilliform (Skin and subcutaneous tissue disorders) | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Rehabilitation therapy (Surgical and medical procedures) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tivozanib Hydrochloride (N=173) | Sorafenib (N=170)
Diarrhoea (Gastrointestinal disorders) | 74 | 91
Stomatitis (Gastrointestinal disorders) | 36 | 38
Nausea (Gastrointestinal disorders) | 51 | 31
Vomiting (Gastrointestinal disorders) | 31 | 25
Abdominal pain (Gastrointestinal disorders) | 21 | 16
Fatigue (General disorders) | 64 | 41
Asthenia (General disorders) | 56 | 40
Hypertension (Vascular disorders) | 73 | 51
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 47 | 16
Decreased appetite (Metabolism and nutrition disorders) | 68 | 51
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 28 | 69
Rash (Skin and subcutaneous tissue disorders) | 17 | 42
Dry skin (Skin and subcutaneous tissue disorders) | 11 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 37
Erythema (Skin and subcutaneous tissue disorders) | 3 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 20
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 11
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 9
Weight decreased (Investigations) | 30 | 37
Blood thyroid stimulating hormone increased (Investigations) | 12 | 2
Dizziness (Nervous system disorders) | 17 | 8
Hypothyroidism (Endocrine disorders) | 31 | 13
Proteinuria (Renal and urinary disorders) | 17 | 6
Oedema peripheral (General disorders) | 16 | 12
Pyrexia (General disorders) | 13 | 18
Abdominal pain upper (Gastrointestinal disorders) | 18 | 12
Constipation (Gastrointestinal disorders) | 19 | 31
Dyspepsia (Gastrointestinal disorders) | 16 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 38 | 26
Back pain (Musculoskeletal and connective tissue disorders) | 32 | 26
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 | 11
Muscle spasms (Musculoskeletal and connective tissue disorders) | 12 | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 12 | 6
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 10
Blood creatinine increased (Investigations) | 13 | 2
Headache (Nervous system disorders) | 20 | 16
Dysgeusia (Nervous system disorders) | 10 | 8
Nasopharyngitis (Infections and infestations) | 12 | 1
Urinary tract infection (Infections and infestations) | 7 | 11
Anaemia (Blood and lymphatic system disorders) | 17 | 23
Hypotension (Vascular disorders) | 9 | 2
Lipase increased (Investigations) | 9 | 4
Aspartate aminotransferase increased (Investigations) | 9 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT02627963/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT02627963/SAP_001.pdf